CLINICAL TRIAL: NCT01261468
Title: Treatment With Spinal Cord Stimulation: Effect on Sensory Parameters
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Danish Pain Research Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: SCS-24h
Record Dates: First submitted 2010-12-15; First posted 2010-12-16 (Estimated); Last update posted 2012-03-15 (Estimated); Status verified 2012-03

CONDITIONS: Chronic Pain
Keywords: Chronic pain; Electric Stimulation Therapy; Neurologic Examination
MeSH Terms: conditions — Chronic Pain

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Active SCS (Active Comparator)
  Interventions: Device: Active SCS
- Inactive SCS (Sham Comparator)
  Interventions: Device: Deactivated

INTERVENTIONS:
Device: Active SCS — SCS IPG activated
  Arms: Active SCS
Device: Deactivated — SCS IPG deactivated
  Arms: Inactive SCS

SUMMARY:
The primary purpose is to study the effect of spinal cord stimulation (SCS) on sensory parameters, using quantitative sensory testing (QST).

Patients with established SCS treatment will be examined with QST. Subjects will be randomized to have their SCS device turned off or kept active (1:1) for a 12-hour period, then be reexamined using the same QST protocol.

After the 2nd examination all patients cross over (ie. inactive devices are activated, active devices are deactivated) and are reexamined after a new 12-hour period.

The investigators expect to demonstrate that SCS treatment has a significant effect on sensory parameters associated with pain hypersensitivity but no significant effect on sensory parameters associated with detection of non-painful stimuli.

ELIGIBILITY:
Inclusion Criteria:

* minimum age 18
* able to understand participant information and cooperate at the neurological examination
* uncomplicated treatment with spinal cord stimulation for at least 3 months
* pain in only one extremity
* treatment effect in only one extremity

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2011-04; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Change in sensory parameters | 24 hours

CONTACTS AND LOCATIONS:
Overall Officials: Troels S Jensen, prof., Study Director — Danish Pain Research Center; Kaare Meier, MD, Principal Investigator — Danish Pain Research Center
Locations (1):
- Danish Pain Research Center, Aarhus C, Denmark

REFERENCES:
- [Background] Kemler MA, Reulen JP, Barendse GA, van Kleef M, de Vet HC, van den Wildenberg FA. Impact of spinal cord stimulation on sensory characteristics in complex regional pain syndrome type I: a randomized trial. Anesthesiology. 2001 Jul;95(1):72-80. doi: 10.1097/00000542-200107000-00016. PMID 11465587